CLINICAL TRIAL: NCT03491150
Title: A Multicenter, Open-Label, Long-Term Extension Of Phase III Studies (BN29552/BN29553) Of Crenezumab In Patients With Alzheimer's Disease
Brief Title: An Open-Label Crenezumab Study in Participants With Alzheimer's Disease
Acronym: CREAD OLE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was discontinued due to an interim analysis in the BN29552 study, which indicated that Crenezumab was unlikely to meet its primary endpoint.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BN40031; 2017-002702-12 (EudraCT Number)
Record Dates: First submitted 2018-03-15; First posted 2018-04-09 (Actual); Results first posted 2020-06-09 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Alzheimer's Disease
Keywords: Dementia; Neurodegenerative Diseases; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurocognitive Disorders; Mental Disorders
MeSH Terms: conditions — Alzheimer Disease; Dementia; Neurodegenerative Diseases; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurocognitive Disorders; Mental Disorders | interventions — crenezumab

STUDY DESIGN:
Intervention Model Description: Open Label Extension (OLE)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Parent Placebo (Placebo Comparator): Participants (who were treated with Placebo in the BN29552/BN29553 Studies) received intravenous (IV) infusion of Crenezumab every 4 weeks (Q4W).
  Interventions: Drug: Crenezumab
- Parent Crenezumab (Experimental): Participants (who were treated with Crenezumab in the BN29552/BN29553 Studies) received intravenous (IV) infusion of Crenezumab every 4 weeks (Q4W).
  Interventions: Drug: Crenezumab

INTERVENTIONS:
Drug: Crenezumab — Crenezumab was administered by intravenous (IV) infusion at 60mg/kg as per the dosing schedule described above.
  Other Names: RO5490245

SUMMARY:
In the BN40031 OLE study, a dose of crenezumab of 60 mg/kg intravenous (IV) every 4 weeks (Q4W) will be offered to all participants who complete Study BN29552 or BN29553 and who meet eligibility criteria in order to evaluate safety in participants on long-term crenezumab treatment and to investigate the effect of crenezumab on the underlying disease process and disease course as an exploratory efficacy objective.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in Study BN29552 or BN29553 and completion of the Week 105 visit.
* Able to provide written informed consent by the patient or legally authorized representative, if required.
* Every effort to have the same caregiver participate throughout the duration of the OLE (Open Label Extension) study who also participated in Study BN29552 or BN29553.
* Willingness and ability to complete all aspects of the study [including MRI (Magnetic Resonance Imaging), lumbar puncture [if applicable], and PET (Positron Emission Tomography) imaging [if applicable].
* Adequate visual and auditory acuity, in the investigator's judgment, sufficient to perform the neuropsychological testing.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a protocol approved contraceptive method and agreement to refrain from donating eggs for at least 8 weeks after last dose.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use a protocol approved contraceptive method for at least 8 weeks after last dose.

Exclusion Criteria:

* Patients who discontinued treatment permanently in Study BN29552 or BN29553 for safety reasons.
* Impaired coagulation.
* Evidence of more than 10 microbleeds and/or ARIA-H (amyloid-related imaging abnormalities-hemosiderin deposition) at the Study BN29552 or BN29553 Week 105 visit, as assessed by central review of MRI.
* Diagnosed with three recurrent, symptomatic ARIA-E (amyloid-related imaging abnormalities-edema/effusion) events or exacerbations of previous events.
* Presence of intracranial lesion that could potentially increase the risk of CNS (Central Nervous System) bleeding.
* At risk of suicide in the opinion of the investigator.
* Alcohol and/or substance abuse or dependence within the past 2 years and during the study.
* Inability to tolerate MRI procedures or contraindication to MRI, including, but not limited to, presence of pacemakers not compatible with MRI, aneurysm clips, artificial heart valves, ear implants, or foreign metal objects in the eyes, skin, or body that would contraindicate an MRI scan; or any other clinical history or examination finding that, in the judgment of the investigator, would pose a potential hazard in combination with MRI.
* Pregnant or lactating, or intending to become pregnant during the study.
* Any other severe or unstable medical condition that, in the opinion of the investigator or Sponsor, could be expected to progress, recur, or change to such an extent that it could put the patient at special risk, bias the assessment of the clinical or mental status of the patient to a significant degree, or interfere with the patient's ability to complete the study assessments.
* Chronic use of anticoagulants or participation in any other investigational drug treatment trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (66):
- United States (32):
  - Shankle Clinic, Newport Beach, California
  - Anderson Clinical Research, Inc., Redlands, California
  - University of California, Davis; Alzheimers Disease Center, Department of Neurology, Sacramento, California
  - UCSF - Memory and Aging Center, San Francisco, California
  - Neurological Research Inst, Santa Monica, California
  - Associated Neurologists PC - Danbury, Danbury, Connecticut
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Yale University School Of Medicine, New Haven, Connecticut
  - Research Center for Clinical Studies, Inc., Norwalk, Connecticut
  - Bradenton Research Center, Bradenton, Florida
  - Brain Matters Research, Inc., Delray Beach, Florida
  - Alzheimer's Research and Treatment Center, Lake Worth, Florida
  - Renstar Medical Research, Ocala, Florida
  - Bioclinica Research, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Stedman Clinical Trials, LLC, Tampa, Florida
  - NeuroStudies.net, LLC, Decatur, Georgia
  - Alexian Brothers Neurosci Inst, Elk Grove Village, Illinois
  - Southern Illinois University, School of Medicine, Springfield, Illinois
  - MidAmerica Neuroscience Institute, Prairie Village, Kansas
  - MMP Neurology, Scarborough, Maine
  - Precise Research Centers, Flowood, Mississippi
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - Advanced Memory Research Institute of NJ, Toms River, New Jersey
  - Behavioral Health Research, Charlotte, North Carolina
  - Guilford Neurologic Associates, Greensboro, North Carolina
  - Oklahoma Clinical Research, Oklahoma City, Oklahoma
  - Summit Research Network Inc., Portland, Oregon
  - Abington Neurological Associates, Willow Grove, Pennsylvania
  - Senior Adults Specialty Research, Austin, Texas
  - Sentara Medical Group, Norfolk, Virginia
  - National Clinical Research Inc.-Richmond, Richmond, Virginia
- Australia (2):
  - Heidelberg Repatriation Hospital; Medical and Cognitive Research Centre, Heidelberg West, Victoria
  - Neurodegenerative Disorders Research; Neurology, West Perth, Western Australia
- Canada (4):
  - Parkwood Hospital; Geriatric Medicine, London, Ontario
  - Kawartha Centre - Redefining Healthy Aging, Peterborough, Ontario
  - The Centre for Memory and Aging, Toronto, Ontario
  - Devonshire Clinical Research Inc., Woodstock, Ontario
- Terveystalo Tampere, Tampere, Finland
- Hopital La Grave; Place Lange, Toulouse Cedec, France
- Klinikum rechts der Isar der TU München; Klinik für Psychiatrie und Psychotherapie, München, Germany
- Prince of Wales Hospital; Dept. of Medicine & Therapeutics, Hong Kong, Hong Kong
- Italy (2):
  - Fondazione Santa Lucia IRCCS, Rome, Lazio
  - Ospedale San Giovanni Calibita Fatebenefratell;Neurologia, Rome, Lazio
- Vilnius University Hospital Santariskiu Clinic, Vilnius, Lithuania
- Mexico (4):
  - Hospital Angeles de Culiacán, Neurociencias Estudios Clínicos SC, Culiacán
  - Hospital Uni; Dr. Jose E. Gonzalez, Monterrey
  - AVIX Investigación Clínica S.C, Monterrey
  - Hospital Universitario de Saltillo, Saltillo
- Centrum Medyczne NeuroProtect, Warsaw, Poland
- Russia (3):
  - State Autonomous Healthcare Institution "Republican Clinical Neurological Center, Kazan'
  - State autonomous institution of healthcare Inter-regional clinical and diagnostic center, Kazan'
  - SHI City Psychoneurological Dispensary #7 (with Hospital), Saint Petersburg
- South Korea (4):
  - Inha University Hospital, Incheon
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
- Spain (6):
  - Fundació ACE, BArcelon, Barcelona
  - Hospital General De Catalunya; Servicio de Neurologia, Sant Cugat del Vallès, Barcelona
  - Hospital Mutua De Terrasa; Servicio de Neurologia, Terrassa, Barcelona
  - Hospital Virgen del Puerto. Servicio de Neurología, Plasencia, Caceres
  - Clinica Universitaria de Navarra; Servicio de Neurología, Pamplona, Navarre
  - Hospital Universitario 12 de Octubre; Servicio de Neurologia, Madrid
- Ondokuz Mayis Univ. Med. Fac.; Neurology, Samsun, Turkey (Türkiye)
- United Kingdom (2):
  - Surrey and Borders NHS Foundation Trust; Research and Development Departmant; Abraham Cowley Unit, Chertsey
  - Charing Cross Hospital, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 66 centers in 16 countries.
Pre-assignment Details: A total of 149 participants were enrolled at 66 centers. These 149 participants represented the Safety Analysis population and data for this population is presented here.
Period: Overall Study
Arm/Group | Parent Placebo | Parent Crenezumab
Started | 76 | 73
Completed | 0 | 0
Not Completed | 76 | 73
Not completed — Adverse Event | 1 | 0
Not completed — Study Terminated by Sponsor | 74 | 70
Not completed — Other | 0 | 1
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Parent Placebo | Parent Crenezumab | Total
Number analyzed (Participants) | 76 | 73 | 149
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.8 (7.6) | 72.0 (7.6) | 72.9 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 38 | 75
  Male | 39 | 35 | 74
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 69 | 69 | 138
  Not Stated | 1 | 1 | 2
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 4 | 2 | 6
  Black or African American | 0 | 1 | 1
  Unknown | 0 | 3 | 3
  White | 72 | 67 | 139

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An Adverse Event is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An adverse event can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events.
Time Frame: Baseline up to 16 weeks after the last dose of study drug (up to 54 weeks).
Population: The Safety analysis population was defined as all participants who consented to the OLE study, including those who enrolled in the OLE but did not receive open-label treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Parent Placebo | Parent Crenezumab
Number analyzed (Participants) | 76 | 73
Percentage of Participants
  AEs | 32.9 | 42.5
  SAEs | 3.9 | 5.5

2. Primary Outcome: Percentage of Participants With Anti-Crenezumab Antibodies
Description: Participants were considered positive or negative for ADA based on their baseline and post-baseline sample results. The number and percentage of participants with confirmed positive ADA levels were determined for Crenezumab and Placebo groups. The prevalence of ADA at baseline was calculated as the proportion of participants with confirmed positive ADA levels at baseline relative to the total number of participants with a sample available at baseline. The incidence of treatment-emergent ADAs was determined as the proportion of participants with confirmed post-baseline positive ADAs relative to the total number of participants that had at least one post-baseline sample available for ADA analysis.
Time Frame: Baseline up to end of study (up to 54 weeks).
Population: Please note that for this Outcome Measure, no Participants were evaluated at all as the existing immunogenicity data from a parent study (Study BN29552) showed a low potential of Crenezumab to induce Anti-Drug Antibodies (ADAs).
Arm/Group | Parent Placebo | Parent Crenezumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 16 weeks after the last dose of study drug (up to 54 weeks).
Arm/Group | Parent Placebo | Parent Crenezumab
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/73
Serious Adverse Events (participants affected / at risk) | 3/76 | 4/73
Other Adverse Events (participants affected / at risk) | 4/76 | 4/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parent Placebo (N=76) | Parent Crenezumab (N=73)
OPTIC ISCHAEMIC NEUROPATHY (Eye disorders) | 0 (0) | 1 (1)
INCARCERATED INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1)
UROSEPSIS (Infections and infestations) | 0 (0) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Parent Placebo (N=76) | Parent Crenezumab (N=73)
FALL (Injury, poisoning and procedural complications) | 4 (5) | 4 (4)

LIMITATIONS AND CAVEATS:
This study was discontinued due to an interim analysis in the BN29552 study, which indicated that Crenezumab was unlikely to meet its primary endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT03491150/Prot_SAP_000.pdf